CLINICAL TRIAL: NCT04530318
Title: Dendritic Cells Therapy Combined With Immunomodulatory Treatment in Multiple Sclerosis
Acronym: TolDecCOMBINEM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Judit Pich (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager. CTU Clinic, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TolDec-COMBINEM; 2020-000737-41 (EudraCT Number)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TolDec (Experimental): Autologous peripheral blood differentiated adult tolerogenic dendritic cells expanded
  Interventions: Other: Autologous peripheral blood differentiated adult tolerogenic dendritic cells expanded
- Placebo (Placebo Comparator): Placebo of dendritic cells
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Autologous peripheral blood differentiated adult tolerogenic dendritic cells expanded — The infusion of the cells / placebo will take place at the Hospital Clínic de Barcelona (weeks 0, 2 and 4).
  Other Names: TolDec
  Arms: TolDec
Other: Placebo — The infusion of the cells / placebo will take place at the Hospital Clínic de Barcelona (weeks 0, 2 and 4).
  Arms: Placebo

SUMMARY:
The aim of this project is to assess properly the clinical efficacy of TolDec therapy by imaging, clinical and surrogate end-points related with the activity of the disease.

DETAILED DESCRIPTION:
Our working hypothesis is to make a combination therapy with low-moderate efficacy immunomodulatory drugs with the aim of increasing efficacy without causing serious adverse effects such as those associated with the available high-efficacy therapies. Cellular therapies represent a highly specific treatment aimed to target selective "pathogenic" cells subsets. Tol-Dec loaded with immunogenic peptides interacts with Ag-specific T lymphocytes inducing regulatory T cells without affecting other cell subsets leading to a antinflammatory shift of immunological responses.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years old.
2. Patients diagnosed with RRMS according to 2017 McDonald criteria.
3. MS disease duration < 10 years.
4. Expanded disability status scale (EDSS) from 0 to < 5.5.
5. Patients eligible to start or already are in on treatment with first line immunomodulatory treatment (interferon beta 1a, interferon beta 1b, glatiramer acetate, teriflunomide or dymethyl-fumarate).
6. Able to sign informed consent.
7. Women of child-bearing potential must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence.

Exclusion Criteria:

1. Presence of a relapse or use of steroids 30 days prior to screening visit.
2. Concomitant use of any type of immunomodulatory / immunosuppressive therapy.
3. Use of previous immunosuppressive or cytotoxic therapy in the last 6 months. Use of previous alemtuzumab, cladribine or bone marrow or stem cell transplant at any time.
4. Patients unable or unwilling to undergo MRI scans.
5. Severe systemic diseases or history of cancer or hereditary familiar cancer.
6. Clinically relevant concomitant disease: cardiac, gastrointestinal, hepatic, pulmonary, neurological, renal or other major disease.
7. Impossibility to proceed to the leukapheresis (e.g. absence of peripheral venous access).
8. Pregnant or breastfeeding women.
9. Drug or alcohol abuse.
10. Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS or to test positive for HIV antibody at screening.
11. Ongoing known bacterial, viral or fungal infection (with the exception of onychomycosis and dermatomycosis), positive hepatitis B surface antigen or hepatitis C antibody tests at screening.
12. Patients with a known history of syphilis or tuberculosis or test positive for syphilis (positive rapid plasma reagin, RPR) or tuberculosis (positive skin test) at screening. Active or latent tuberculosis (TB).
13. Dementia or severe psychiatric, cognitive or behavioral problems or other comorbidity that may interfere with the compliance to the protocol.
14. Any other clinically relevant medical or surgical condition, which, in the opinion of the investigator, would put the subject at risk by participating in the study.
15. Participation in other experimental studies within the previous 90 days prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the number of CUA lesion (mean number of the sum at week 12, 18 and 24). | week 12, 18 and 24
Proportion of patients with any Grade 3 -4 adverse events related to product administration during the study period. | week 24
Proportion of patients with any Grade 3 -4 adverse events related to study product. | week 24

SECONDARY OUTCOMES:
Proportion of patients with any Grade 3 -4 adverse events related to study product. | week 24
Proportion of patients with any SAE events related to study product. | week 24
Proportion of patients with at least one MS relapse during the study period. | week 24
Total number of MS relapse at 24 weeks. | week 24
Time to first MS relapse during the study period. | week 24
Changes from baseline in the disability progression by Expanded Disability Status Scale (EDSS) at week 24. | week 24
Changes from baseline in the disability progression by Multiple Sclerosis Functional Composite (MSFC) at week 24. | week 24
Changes from baseline in the number of CUA lesion at week 24. | week 24
Proportion of patients free from CUA lesion, gadolinium-enhancing lesions on T1 MRI and new or enlarged lesions on T2-MRI thought the 24 weeks of study. | week 24
Changes from baseline in the number of Gd-enhancing T1 lesions by scan (mean number of the sum at week 12, 18 and 24) and at week 24. | week 24
Changes from baseline in number of new or enlarging T2 lesions by scan (mean number of the sum at week 12, 18 and 24) and at week 24. | week 24
Changes from baseline in brain global, white and gray matter volume and cervical cord volume on MRI at 24 weeks. | week 24
Changes from baseline in the number of cortical lesions on MRI at 24 weeks. | week 24
Changes from baseline in MR measurements of diffuse damage of brain tissue by MTR at 24 weeks | week 24
Changes from baseline in MR measurements of relaxation times of T1 and T2 by MTR at 24 weeks. | week 24
Changes in DTI measures as mean diffusivity (MD), fractional anisotropy (FA), radial diffusivity (Dr) and axial diffusivity (Da) at 24 weeks. | week 24
Changes from baseline in cytokine production (including IFNgamma, IL-17, IL-4 and IL-10) in response to specific peptide stimulation in peripheral blood mononuclear cells (PBMCs) culture supernatants at 12 and 24 weeks. | week 24
Changes from baseline in T cell proliferation to immunogenic peptides at 12 and 24 weeks. | week 24
Changes from baseline in immune cell subsets in PBMCs including PBMC subtypes, T lymphocytes subpopulations and Treg subsets, CD4 and CD8 GM-CSF 'encephalitogenic' T cells and T cell subtypes by activation memory phenotype at 12 and 24 weeks. | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Blanco, MD, Study Chair — Hospital Clinic of Barcelona
Locations (5):
- Spain (5):
  - Hospital Moisés Broggi, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No